CLINICAL TRIAL: NCT06448416
Title: Assessment of Unilateral Biportal Endoscopy Technique Applied to Treatment of Degenerative Lumbar Pathologies
Acronym: UBEVAL
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: RGDS-2023-12-014
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unilateral Biportal Endoscopy (UBE) Technique: Patient with LDH treated by UBE
  Interventions: Procedure: UBE

INTERVENTIONS:
Procedure: UBE — Patients with HDL were treated with UBE

SUMMARY:
Lumbar disc herniation (HDL) is one of the main causes for low back pain and sciatica. Although non surgical care remains the gold standard as first treatment, lumbar discectomy is used to effectively relieve symptoms that persist for prolonged periods.

With surgical techniques evolution, minimally invasive spine surgery has emerged in recent decades as an alternative to conventional open surgery and is widely used for HDL treatment. Several minimally invasive surgical endoscopic techniques have been developed for disc herniation: Single Portal Endoscopy (SE), Video Assisted Endoscopic Discectomy, and recently Unilateral Biportal Endoscopy (UBE).

Currently, SE is considered as the minimally invasive surgery gold standard for HDL but, over the past two years, UBE for the treatment of degenerative lumbar diseases has increased exponentially with faster learning curve than other endoscopic techniques.

As an emerging technique, further studies are needed to better understand UBE. This is why Dr. Cristini's team wish to analyze a cohort of patients for whom this technique has been used since July 2022, in particular the complication rate.

Controlling a new technique requires a learning phase. This is why Dr. Cristini's team also wishes to describe the learning curve on the cohort of patients for whom UBE was used since July 2022.

DETAILED DESCRIPTION:
Lumbar disc herniation (HDL) is one of the main causes for low back pain and sciatica, affecting 1 to 5% of the population each year. Although non surgical care remains the gold standard as first treatment, lumbar discectomy is used to effectively relieve symptoms that persist for prolonged periods.

With surgical techniques evolution, minimally invasive spine surgery has emerged in recent decades as an alternative to conventional open surgery and is widely used for HDL treatment. Compared to traditional open surgery, minimally invasive surgical technique offers muscle and bone sparing, pain reduction and faster recovery, allowing patient management in Enhanced Recovery After Surgery (RAAC).

Several minimally invasive surgical endoscopic techniques have been developed for disc herniation: Single Portal Endoscopy (SE), Video Assisted Endoscopic Discectomy, and recently Unilateral Biportal Endoscopy (UBE). SE relies on a single entry route whereas UBE is based on two entry routes : one way for optical instruments and saline irrigation system and one way for surgical instruments. Currently, SE is considered as the minimally invasive surgery gold standard for HDL treatment thanks to its advantages for controlling muscles trauma, reducing hospital stay and maintaining spinal segment stability.

Over the past two years, UBE for the treatment of degenerative lumbar diseases has increased exponentially with faster learning curve than other endoscopic techniques.

UBE allows a wider field of vision, wide and ergonomic operating gestures, is minimally invasive and contributes to complete nervous decompression and faster recovery. With UBE, the surgeon can use one hand to guide endoscope and he other one to guide surgical instruments . In addition, UBE generates less trauma, less bleeding, rapid recovery and good effectiveness in HDL treatment . UBE can significantly reduce postoperative nerve fibrosis, and postoperative spinal instability incidence.

During UBE, some postoperative complications have been described as poor treatment effectiveness (nucleus pulposus nucleus residue), epidural hematoma, dural tear, nerve root injury and incomplete surgery.

As an emerging technique, further studies are needed to better understand UBE. This is why Dr. Cristini's team wish to analyze a cohort of patients for whom this technique has been used since July 2022, in particular the complication rate.

Controlling a new technique requires a learning phase. Chen, L et al. showed that the operation duration and the postoperative hospitalization duration, were reduced from the 24th patient until the 97th patient out of a cohort of 97 patients with lumbar disc herniation treated by UBE. However, there was no significant difference in the visual analogue scale (VAS) and the Oswestry disability index (ODI) in all operated patients. This indicates that UBE still guarantees clinical effect and safety on all operated patients. This is why Dr. Cristini's team also wishes to describe the learning curve on the cohort of patients for whom UBE was used since July 2022.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years old
* Patient with lumbar disc herniation or non-instrumented degenerative lumbar pathology
* Patient operated with UBE technique

Exclusion Criteria:

* Patient with extreme lateral disc herniation.
* Patient suffering from other serious illnesses
* Patient with lumbar instability, lumbar infection or lumbar tumor,
* Patient with multi-segmental lumbar disease requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population means patients who fulfill inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Patient complication rate | 2 days
  Complications will include epidural hematoma, nerve root injury, neurological deficit, dural breach or tear, incomplete surgery, epileptic crisis, hypothermia. Other complications will be HDL recurrence, pain neuropathy, infection and thromboembolic complications

SECONDARY OUTCOMES:
surgeon learning curve | 21 months
  UBE learning curve will be assessed with surgery time (minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital CLAIRVAL, Marseille, France

IPD SHARING:
Plan to Share IPD: No